CLINICAL TRIAL: NCT00787007
Title: Randomized, Double-Blind, Single Rising Dose Study of S-equol in Normal Volunteers
Brief Title: Safety and Pharmacokinetic Study of S-Equol in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ausio Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: AUS-CT01
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
Keywords: healthy volunteers; pharmacokinetics
MeSH Terms: interventions — Equol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- 1 (Experimental): 10 mg
  Interventions: Drug: S-equol
- 2 (Experimental): 20 mg, fasted and fed
  Interventions: Drug: S-equol
- 3 (Experimental): 40 mg
  Interventions: Drug: S-equol
- 4 (Experimental): 80 mg
  Interventions: Drug: S-equol
- 5 (Experimental): 160 mg
  Interventions: Drug: S-equol
- 6 (Experimental): 320 mg
  Interventions: Drug: S-equol
- 7 (Placebo Comparator): placebo capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S-equol — capsule, oral, single dose
  Other Names: AUS-131
  Arms: 1; 2; 3; 4; 5; 6
Drug: Placebo — capsule, oral, single dose
  Arms: 7

SUMMARY:
The purpose of this study is 1) to test the safety of S-equol in healthy volunteers and 2) to see how quickly S-equol enters the bloodstream, is distributed in the body, and broken down and removed, when taken with food or without food.

DETAILED DESCRIPTION:
The study is a double blind, randomized, placebo-controlled, dose-escalation study of the safety and tolerability of single doses of S-equol up to 320 mg in healthy male and female adult subjects. Approximately 8 qualified volunteers will be selected at each dose level and randomly assigned to receive S-equol or placebo, in the fasted state. For the 20 mg dose group, subjects will complete two treatment periods, one in the fasted state, and one in the fed state.

A safety review of study results for each dose group will occur when Day 8 follow-up visit safety data are available, and prior to enrollment/dosing of the next subsequent dose group. Given favorable safety review of a dose group's experience, the subsequent dose group will be enrolled/dosed at least 10 days after the previous group's dosing.

Pharmacokinetic evaluations consist of determination of plasma and urine concentrations of free and total conjugated S-equol at various time points. Safety evaluations include physical examination,vital signs, ECG, serum chemistry, hematology, and urinalysis, 12-lead telemetry, and assessment of clinical signs and symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers aged 18 to 65 years, inclusive
* Female subjects must be non-pregnant and non-lactating; surgically sterile, post-menopausal or be using an acceptable non-hormonal method of birth control
* Must not have used any hormonal agents or devices within 4 weeks prior to enrollment
* In good health as determined by a physician
* BMI between 18 and 30, inclusive
* Normal clinical laboratory test results
* Negative drug and alcohol toxicology screens
* Negative HIV antibody and hepatitis panel screening results
* For men over 44 years of age, PSA ≤ 2.0 ng/mL
* For women over 44 years of age, normal mammography and pelvic ultrasound
* Protein C and Protein S activity levels above the lower limit of normal
* Negative for Factor V Leiden.

Exclusion Criteria:

* History of any chronic, subacute or acute condition of clinical significance
* Total bilirubin level >0.9, conjugated bilirubin >0.4, or unconjugated bilirubin >0.8
* Fasting cholesterol level >280 mg/dL; fasting triglyceride level >1.5 x ULN
* History of thromboembolic events or estrogen-dependent benign or malignant neoplasm
* Resting systolic blood pressure >140 mm Hg or <90 mm Hg, or diastolic blood pressure >90 mm Hg or <60 mm Hg
* Resting pulse >100 beats/minute or <45 beats/minute
* Abnormal 12-lead ECG or telemetry results
* Subject is unwilling or unable to comply with study rules
* History of sudden cardiac death in the immediate family, or a personal history of cardiac disease, treated hypertension, congestive heart failure, or unexplained syncope
* History of cancer, other than basal cell carcinoma or stage 1 squamous cell carcinoma, that has not been successfully treated
* Use of any prescription or over-the-counter medication within 1 week prior to Day -1 or anticipates the need for any medication during the course of the study
* History or intolerance to estrogen medication
* History of substance abuse, drug addiction, or alcoholism within 3 years
* Inability to abstain from alcohol, caffeine, Yerba mate tea, or from grapefruit, grapefruit juice or flavonoid-rich foods from 48 hours prior to the administration of study medication and throughout the duration of the study.
* History of smoking or any use of a tobacco or nicotine containing product within 6 months
* Donated blood or blood products within 30 days
* Mental instability or inability to be compliant with the protocol
* Subject has received an investigational test substance within 60 days or anticipates receiving any investigational test substance other than S-equol during the course of this study
* Subject has been previously enrolled in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of ascending, single oral doses of S-equol, administered in fasted and fed states, in healthy male and female volunteers. | Continuous

SECONDARY OUTCOMES:
To evaluate the single dose pK profile of S-equol in the fed and fasted state. To compare the pK profiles of younger and older and male and female volunteers. | Variable

CONTACTS AND LOCATIONS:
Locations (1):
- Charles River, Tacoma, Washington, United States